CLINICAL TRIAL: NCT02166502
Title: Nevirapine Dosing in Neonates for Prophylaxis of Mother-to-Child-Transmission (MTCT) of HIV Infection
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Foundation for AIDS Research (CANFAR) (Other); Children's Hospital of Eastern Ontario (Other); Unity Health Toronto (Other); Mount Sinai Hospital, Canada (Other)
Responsible Party: Principal Investigator, Ari Bitnun, Staff Physician, The Hospital for Sick Children
Other Study IDs: 1000029134
Record Dates: First submitted 2014-06-05; First posted 2014-06-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Human Immunodeficiency Virus; HIV; Vertical Infection Transmission
Keywords: pediatric; HIV; prevention; prophylaxis; nevirapine
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nevirapine: The patients in this study are newborn infants clinically prescribed combination antiretroviral treatment with nevirapine for prevention of mother-to-child HIV transmission.

SUMMARY:
The purpose of this study is to determine whether the current dose of nevirapine recommended in the Ontario Ministry of Health vertical transmission prevention protocol achieves therapeutic drug levels in newborn infants at high risk of HIV infection.

DETAILED DESCRIPTION:
Although nevirapine (NVP) is often given as part of combination antiretroviral therapy (cART) at our institutions for prevention of vertical transmission (VT) in high risk infants, the optimal prophylactic dose of nevirapine is unknown. The National Institute of Health (NIH) guidelines currently recommend a single 2 mg/kg dose of nevirapine given to the infant within 72 hours of birth, however, this dose is not being used in practice given the controversies previously described with single-dose nevirapine. In the absence of any guidance to inform the multiple daily dosing of nevirapine for prophylaxis of VT, we are currently using the treatment dose for infants >15 days of age of 150 mg/m2 once daily for 14 days, then increasing to 150 mg/m2 twice daily for 14 days. This is analogous to the treatment dosing of triple antiretrovirals (ARVs) that is given for occupational post-exposure prophylaxis. Nevirapine is given for 4 weeks total with zidovudine (AZT) and lamivudine (3TC), followed by 2 additional weeks of AZT and 3TC to prevent the development of nevirapine resistance from its long half life. Stopping all 3 drugs simultaneously would result in a period of functional NVP monotherapy, resulting in a risk of NVP resistance should the infant become infected despite prophylaxis. Since the dose of nevirapine being used in our clinic populations for prevention of VT is higher than has been previously studied in neonates, it is important to evaluate the safety and efficacy of this dosing regimen, using therapeutic drug monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants prescribed combination antiretroviral treatment with nevirapine for prevention of mother-to-child HIV transmission. These infants are routinely referred to the Hospital for Sick Children (SickKids) and Children's Hospital of Eastern Ontario (CHEO) HIV clinics in Toronto and Ottawa, respectively, for ongoing management. The majority of referrals are from Mount Sinai Hospital and St. Michael's Hospital in Toronto, and the Ottawa General Hospital in Ottawa.
* Voluntary informed consent by the legal guardian

Exclusion Criteria:

* Infants born prior to 32 weeks gestational age;
* Infants with life-threatening medical conditions;
* Infants unable to take oral medication;
* Infants born to women considered at high risk of harboring nevirapine resistance mutations in whom Kaletra (lopinavir/ritonavir) is a therapeutic option (e.g. term neonates) will be excluded and prescribed Kaletra rather than nevirapine

Max Age: 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The patients in this study are newborn infants clinically prescribed combination antiretroviral treatment with nevirapine for prevention of mother-to-child HIV transmission. These infants are routinely referred to the SickKids and CHEO HIV clinics in Toronto and Ottawa, respectively, for ongoing management. The majority of referrals are from Mount Sinai Hospital and St. Michael's Hospital in Toronto, and the Ottawa General Hospital in Ottawa.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2012-02; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of nevirapine trough (Cmin) plasma levels that are above or below the target range for prophylaxis | Weeks 1, 2, and 4

SECONDARY OUTCOMES:
Final dose of nevirapine | Week 4
  Final dose of nevirapine required to achieve target plasma trough concentrations at week 4
Derived pharmacokinetic parameters | Week 4
  Derived pharmacokinetic parameters volume of distribution (Vd)(L/kg), elimination rate (ke), clearance (mL/kg/hr), Cmin (ug/L), Cmax (ug/L), Tmax (hrs), and Area under the Curve (AUC)
Association between nevirapine levels and incidence of adverse effects | Weeks 1, 2 and 4
  Number of adverse events among patients with therapeutic vs. supratherapeutic nevirapine levels
Association between patient characteristics and differences in nevirapine levels | Baseline, Week 1, 2 and 4
  Patient characteristics that may explain differences in nevirapine levels including chronologic and gestational age, weight, and ethnic background.
Rate of vertical transmission of HIV | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ari Bitnun, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario